CLINICAL TRIAL: NCT06782100
Title: MRI Guided Management of Occlusive Peripheral Arterial Disease
Status: Recruiting | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Triisha Roy, Vascular Surgeon- Scientist, The Methodist Hospital Research Institute
Other Study IDs: PRO00027258; R01HL174587 (NIH)
Record Dates: First submitted 2024-12-16; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Vascular Diseases
Keywords: MRI Guided Management of Occlusive Peripheral Arterial Disease; PAD; Peripheral Vascular Disease; PVI; MRI; MRA
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood vessel samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Amputation Arm: In an ex vivo human cadaveric model, post-PVI histopathologic analysis will be used to uncover the impact of plaque type on device safety (POBA versus atherectomy) and performance, facilitating evidence-based device selection to mitigate complications. Using a randomized approach, the investigator will compare plain balloon angioplasty to orbital atherectomy prior to angioplasty in amputated legs from PAD patients with plaques characterized into 4 categories based their MRI-histology: concentric calcium, eccentric calcium, fibrous plaque, and soft plaques (smooth muscle and thrombus).
- Revascularization Arm: Patient Imaging Protocol: Scans will be performed on 100 patients enrolled into the study population using a 3T MAGNETOM scanner (Siemens) at the Houston Methodist Research Institute Translational Imaging Center. The investigator will use pre-operative images captured using the optimized MRI-histology sequences to score lesions. Physicians performing PVI will be blinded to the pre-operative MRI-histology images and anatomic scores and will make treatment decisions based on their standard of care. The investigator expect MRI-histology plaque scores predict which patients will have PVI failures due to untraversable plaque, and it may also foresee the potential need of adjunctive devices or alternative approaches for successful PVI

SUMMARY:
The goal of this observational study is to identify which plaque lesions in patients with peripheral arterial disease are impenetrable and to determine which devices minimize vessel wall injury.

Patients undergoing intervention will have an MRI scan prior to their planned percutaneous vascular intervention to assess the plaque and predict procedural difficulty.

Patients undergoing lower limb amputation due to peripheral arterial disease will have their limbs included into a second arm of the study The limb will undergo an MRI scan to assess the plaque. The investigator will then test two different devices and assess the effects of these devices on the vessel wall.

DETAILED DESCRIPTION:
Please see attached study protocol.

ELIGIBILITY:
Inclusion Criteria:

A. General Inclusion Criteria:

i. All patients will be ≥ 40 years old with PAD (Rutherford Category 4, 5, 6)

B. Anatomic inclusion criteria:

i. At least 1 target lesion below-the-knee in native vessels in one or both limbs ii. Target lesion reference vessel diameter between 2.0 - 4.0 mm by investigator visual estimate iii. Target lesion with > 50% stenosis by investigator visual estimate

Exclusion Criteria:

A. General Exclusion Criteria:

i. Rutherford category 0, 1, 2, 3 of target limb, Failure or refusal to provide written informed consent, MRI Contraindications

B. Anatomic Exclusion Criteria:

ii. Aim 2 only - Chronic total occlusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For Revascularization Arm: Patients will be enrolled from Vascular surgical Care at Houston Methodist Hospital and undergoing lower limb PVI.
  For Amputation Arm: Patients undergoing Major lower limb amputation at Houston Methodist Hospital with PAD.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Patient primary Outcome | Intraprocedural - the outcome is at the time of the procedure, it is not a follow up outcome.
  PVI failure due to inability to cross the target plaque with a guidewire.
Amputation Arm Outcome | From Experiment and detected during Histological Evaluation (there is no timeframe from this as it is after the experiment on histological analysis)
  Presence of dissections on histology (number of dissections i.e. count, idissection score)

SECONDARY OUTCOMES:
Patient outcome measures | Intraprocedural
  1. Plaque-crossing time (seconds),
  2. successful target lesion revascularization (yes or no)
  3. use of adjunct devices beyond plain balloon angioplasty (record name of device[s])
  4. injury/dissection of vessel requiring stent (record event title e.g. dissection)
  5. plaque embolization (yes/no)
  6. number and stiffness of wires and catheters used (record device names)
  7. subintimal crossing (yes/no)
  8. outcomes after antegrade/retrograde access (successful/unsuccessful)
Amputation Arm Outcomes | From Experiment and Histologicla Examination
  1. Minimal inflation pressure
  2. mean luminal gain percentage based on IVUS
  3. severity of dissections using iDissection classification and
  4. endothelial injury
Patient Outcome Measure | Intraprocedural
  Hypothesis: Women will have less MRI-defined hard lesions and plaques that are easier to cross Comparison Groups: Women vs. Men Primary Outcome: PVI failure due to inability to cross the target plaque with a guidewire (record number of hard lesions i.e. count, comparing men and women)

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Based on ethical and legal considerations, only the following data produced in the course of the project will be preserved and shared on a data repository platform: MRI, angiography, Cone Beam CT, and histology data.The final dataset will include self-reported demographic data. We will share de-identified individualparticipant level (IPD) data. Appropriate measures such as assigning a random code to each participant will be used for data de-identification and sharing, and informed consent forms will reflect those plans.

REFERENCES:
- [Background] Csore J, Karmonik C, Wilhoit K, Buckner L, Roy TL. Automatic Classification of Magnetic Resonance Histology of Peripheral Arterial Chronic Total Occlusions Using a Variational Autoencoder: A Feasibility Study. Diagnostics (Basel). 2023 May 31;13(11):1925. doi: 10.3390/diagnostics13111925. PMID 37296778
- [Background] Barisano G, Sepehrband F, Ma S, Jann K, Cabeen R, Wang DJ, Toga AW, Law M. Clinical 7 T MRI: Are we there yet? A review about magnetic resonance imaging at ultra-high field. Br J Radiol. 2019 Feb;92(1094):20180492. doi: 10.1259/bjr.20180492. Epub 2018 Nov 1. PMID 30359093
- [Background] Shammas NW, Shammas WJ, Jones-Miller S, Torey JT, Armstrong EJ, Radaideh Q, Shammas GA. Optimal Vessel Sizing and Understanding Dissections in Infrapopliteal Interventions: Data From the iDissection Below the Knee Study. J Endovasc Ther. 2020 Aug;27(4):575-580. doi: 10.1177/1526602820924815. Epub 2020 May 18. PMID 32419593
- [Background] Horie K, Tanaka A, Taguri M, Kato S, Inoue N. Impact of Prolonged Inflation Times During Plain Balloon Angioplasty on Angiographic Dissection in Femoropopliteal Lesions. J Endovasc Ther. 2018 Dec;25(6):683-691. doi: 10.1177/1526602818799733. Epub 2018 Sep 11. PMID 30203701
- [Background] Ebisawa S, Kohsaka S, Muramatsu T, Kashima Y, Okamura A, Yamane M, Sakurada M, Matsuno S, Kijima M, Habara M. Derivation and validation of the J-CTO extension score for pre-procedural prediction of major adverse cardiac and cerebrovascular events in patients with chronic total occlusions. PLoS One. 2020 Sep 11;15(9):e0238640. doi: 10.1371/journal.pone.0238640. eCollection 2020. PMID 32915843
- [Background] Werncke T, Ringe KI, von Falck C, Kruschewski M, Wacker F, Meyer BC. Diagnostic confidence of run-off CT-angiography as the primary diagnostic imaging modality in patients presenting with acute or chronic peripheral arterial disease. PLoS One. 2015 Apr 2;10(3):e0119900. doi: 10.1371/journal.pone.0119900. eCollection 2015. PMID 25835948
- [Background] Mohebali J, Patel VI, Romero JM, Hannon KM, Jaff MR, Cambria RP, LaMuraglia GM. Acoustic shadowing impairs accurate characterization of stenosis in carotid ultrasound examinations. J Vasc Surg. 2015 Nov;62(5):1236-44. doi: 10.1016/j.jvs.2015.06.137. PMID 26506272
- [Background] Roy T, Liu G, Shaikh N, Dueck AD, Wright GA. Puncturing Plaques. J Endovasc Ther. 2017 Feb;24(1):35-46. doi: 10.1177/1526602816671135. Epub 2016 Sep 25. PMID 27659155
- [Background] Ebert MLA, Schmidt VF, Pfaff L, von Thaden A, Kimm MA, Wildgruber M. Animal Models of Neointimal Hyperplasia and Restenosis: Species-Specific Differences and Implications for Translational Research. JACC Basic Transl Sci. 2021 Aug 11;6(11):900-917. doi: 10.1016/j.jacbts.2021.06.006. eCollection 2021 Nov. PMID 34869956
- [Background] Hsu CC, Kwan GN, Singh D, Rophael JA, Anthony C, van Driel ML. Angioplasty versus stenting for infrapopliteal arterial lesions in chronic limb-threatening ischaemia. Cochrane Database Syst Rev. 2018 Dec 8;12(12):CD009195. doi: 10.1002/14651858.CD009195.pub2. PMID 30536919
- [Background] Jones DW, Schanzer A, Zhao Y, MacKenzie TA, Nolan BW, Conte MS, Goodney PP; Vascular Study Group of New England. Growing impact of restenosis on the surgical treatment of peripheral arterial disease. J Am Heart Assoc. 2013 Nov 25;2(6):e000345. doi: 10.1161/JAHA.113.000345. PMID 24275626
- [Background] Nolan BW, De Martino RR, Stone DH, Schanzer A, Goodney PP, Walsh DW, Cronenwett JL; Vascular Study Group of New England. Prior failed ipsilateral percutaneous endovascular intervention in patients with critical limb ischemia predicts poor outcome after lower extremity bypass. J Vasc Surg. 2011 Sep;54(3):730-5; discussion 735-6. doi: 10.1016/j.jvs.2011.03.236. Epub 2011 Jul 29. PMID 21802888
- [Background] Roy TL, Chen HJ, Dueck AD, Wright GA. Magnetic resonance imaging characteristics of lesions relate to the difficulty of peripheral arterial endovascular procedures. J Vasc Surg. 2018 Jun;67(6):1844-1854.e2. doi: 10.1016/j.jvs.2017.09.034. Epub 2017 Dec 13. PMID 29248239
- [Background] Bradbury AW, Moakes CA, Popplewell M, Meecham L, Bate GR, Kelly L, Chetter I, Diamantopoulos A, Ganeshan A, Hall J, Hobbs S, Houlind K, Jarrett H, Lockyer S, Malmstedt J, Patel JV, Patel S, Rashid ST, Saratzis A, Slinn G, Scott DJA, Zayed H, Deeks JJ; BASIL-2 Investigators. A vein bypass first versus a best endovascular treatment first revascularisation strategy for patients with chronic limb threatening ischaemia who required an infra-popliteal, with or without an additional more proximal infra-inguinal revascularisation procedure to restore limb perfusion (BASIL-2): an open-label, randomised, multicentre, phase 3 trial. Lancet. 2023 May 27;401(10390):1798-1809. doi: 10.1016/S0140-6736(23)00462-2. Epub 2023 Apr 25. PMID 37116524
- [Background] Kristensen MT, Holm G, Kirketerp-Moller K, Krasheninnikoff M, Gebuhr P. Very low survival rates after non-traumatic lower limb amputation in a consecutive series: what to do? Interact Cardiovasc Thorac Surg. 2012 May;14(5):543-7. doi: 10.1093/icvts/ivr075. Epub 2012 Jan 31. PMID 22298857
- [Background] Misra S, Shishehbor MH, Takahashi EA, Aronow HD, Brewster LP, Bunte MC, Kim ESH, Lindner JR, Rich K; American Heart Association Council on Peripheral Vascular Disease; Council on Clinical Cardiology; and Council on Cardiovascular and Stroke Nursing. Perfusion Assessment in Critical Limb Ischemia: Principles for Understanding and the Development of Evidence and Evaluation of Devices: A Scientific Statement From the American Heart Association. Circulation. 2019 Sep 17;140(12):e657-e672. doi: 10.1161/CIR.0000000000000708. Epub 2019 Aug 12. PMID 31401843
- [Background] Criqui MH, Matsushita K, Aboyans V, Hess CN, Hicks CW, Kwan TW, McDermott MM, Misra S, Ujueta F; American Heart Association Council on Epidemiology and Prevention; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Lifestyle and Cardiometabolic Health; Council on Peripheral Vascular Disease; and Stroke Council. Lower Extremity Peripheral Artery Disease: Contemporary Epidemiology, Management Gaps, and Future Directions: A Scientific Statement From the American Heart Association. Circulation. 2021 Aug 31;144(9):e171-e191. doi: 10.1161/CIR.0000000000001005. Epub 2021 Jul 28. PMID 34315230
- [Background] Creager MA, Matsushita K, Arya S, Beckman JA, Duval S, Goodney PP, Gutierrez JAT, Kaufman JA, Joynt Maddox KE, Pollak AW, Pradhan AD, Whitsel LP. Reducing Nontraumatic Lower-Extremity Amputations by 20% by 2030: Time to Get to Our Feet: A Policy Statement From the American Heart Association. Circulation. 2021 Apr 27;143(17):e875-e891. doi: 10.1161/CIR.0000000000000967. Epub 2021 Mar 25. PMID 33761757
- [Background] Zia S, Juneja A, Shams S, Faheem B, Shariff MA, Singh K, Schor J, Deitch J. Contemporary outcomes of infrapopliteal atherectomy with angioplasty versus balloon angioplasty alone for critical limb ischemia. J Vasc Surg. 2020 Jun;71(6):2056-2064. doi: 10.1016/j.jvs.2019.08.254. Epub 2019 Nov 11. PMID 31727459
- [Background] Farber A, Menard MT, Conte MS, Kaufman JA, Powell RJ, Choudhry NK, Hamza TH, Assmann SF, Creager MA, Cziraky MJ, Dake MD, Jaff MR, Reid D, Siami FS, Sopko G, White CJ, van Over M, Strong MB, Villarreal MF, McKean M, Azene E, Azarbal A, Barleben A, Chew DK, Clavijo LC, Douville Y, Findeiss L, Garg N, Gasper W, Giles KA, Goodney PP, Hawkins BM, Herman CR, Kalish JA, Koopmann MC, Laskowski IA, Mena-Hurtado C, Motaganahalli R, Rowe VL, Schanzer A, Schneider PA, Siracuse JJ, Venermo M, Rosenfield K; BEST-CLI Investigators. Surgery or Endovascular Therapy for Chronic Limb-Threatening Ischemia. N Engl J Med. 2022 Dec 22;387(25):2305-2316. doi: 10.1056/NEJMoa2207899. Epub 2022 Nov 7. PMID 36342173
- [Background] Boulton AJ, Vileikyte L, Ragnarson-Tennvall G, Apelqvist J. The global burden of diabetic foot disease. Lancet. 2005 Nov 12;366(9498):1719-24. doi: 10.1016/S0140-6736(05)67698-2. PMID 16291066